CLINICAL TRIAL: NCT03117387
Title: Evaluation of the Tof Cuff for Perioperative Neuromuscular Transmission Monitoring During Recovery of Moderate and Deep Neuromuscular Block Compared to Acceleromyography and Electromyography
Brief Title: Evaluation of the Tof Cuff for Perioperative Neuromuscular Transmission
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Albert Dahan, MD PhD, Leiden University Medical Center
Other Study IDs: P17.050
Record Dates: First submitted 2017-03-28; First posted 2017-04-17 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-09

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- moderate neuromuscular block, normal body mass index: Patients with normal BMI (< 30) who will receive a moderate neuromuscular block (train of four 1-3 twitches)
  Interventions: Diagnostic Test: Measurements of the level of neuromuscular blockade
- deep neuromuscular block, normal body mass index: Patients with normal BMI (< 30) who will receive a deep neuromuscular block (post tetanic count of 1-2 twitches)
  Interventions: Diagnostic Test: Measurements of the level of neuromuscular blockade
- moderate neuromuscular block, high body mass index: Patients with high BMI (> 30) who will receive a moderate neuromuscular block (train of four 1-3 twitches)
  Interventions: Diagnostic Test: Measurements of the level of neuromuscular blockade
- deep neuromuscular block, high body mass index: Patients with high BMI (> 30) who will receive a deep neuromuscular block (post tetanic count of 1-2 twitches)
  Interventions: Diagnostic Test: Measurements of the level of neuromuscular blockade

INTERVENTIONS:
Diagnostic Test: Measurements of the level of neuromuscular blockade — Study participant were not prospectively exposed to an intervention. Administration of a moderate or deep neuromuscular blockade is at the discretion of the attending anesthesiologist. Study participants only received diagnostic non-invasive monitoring. In routine clinical care the neuromuscular blockade is monitored non-invasively by either acceleromyography, electromyography or by the TOF-Cuff. In this study participants were monitored by the monitors and were not exposed to any additional risk and no effect of an intervention was assessed in this study.

SUMMARY:
Acceleromyography (AMG) is the most wide spread used method to assess neuromuscular block during anesthesia. However AMG is known to be inaccurate when compared to the gold standard in neuromuscular transmission monitoring, electromyography (EMG). Furthermore when the patients arms require to be positioned next to the body and beneath surgical drapes, AMG measurements are often hindered and inaccurate. The TOF cuff is a new device which measures neuromuscular blockade at the upper arm with a blood pressure cuff. It overcomes the previously mentioned disadvantages of AMG. However, it validity compared to EMG and AMG has not yet fully been investigated.

This study aims to compare the bias, limits of agreement and precision of the Train-of-Four cuff relative to AMG and EMG during recovery of moderate and deep neuromuscular block in patients with normal body mass index and morbidly obese patients.

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesiologist Physical Status class I-III
* >18 years of age
* Ability to give oral and written informed consent

Exclusion Criteria:

* Known or suspected neuromuscular disorders impairing neuromuscular function;
* Allergies to muscle relaxants, anesthetics or narcotics;
* A (family) history of malignant hyperthermia;
* Women who are or may be pregnant or are currently breast feeding;
* Renal insufficiency, as defined by a glomerular filtration rate < 30 ml/min
* Scheduled for anesthesia without the use of muscle relaxants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: American society of Anesthesiologist Physical Status class I-III patients >18 years of age BMI either < 30 or > 30 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Medisch Centrum Haaglanden / Nederlandse Obesitas Kliniek, The Hague, South Holland

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Neuromuscular Block, Normal Body Mass Index: Patients with normal normal body mass index(< 30) who will receive a moderate neuromuscular block (train of four 1-3 twitches) as determined by the attending anesthesiologist.
  The TOF-Cuff was compared with electromyography
- Deep Neuromuscular Block, Normal Body Mass Index: Patients with normal normal body mass index(< 30) who will receive a deep neuromuscular block (post tetanic count of 1-2 twitches) as determined by the attending anesthesiologist.
  The TOF-Cuff was compared with electromyography
- Moderate Neuromuscular Block, High Body Mass Index: Patients with high normal body mass index(> 30) who will receive a moderate neuromuscular block (train of four 1-3 twitches) as determined by the attending anesthesiologist.
  The TOF-Cuff was compared with electromyography
- Deep Neuromuscular Block, High Body Mass Index: Patients with high normal body mass index(> 30) who will receive a deep neuromuscular block (post tetanic count of 1-2 twitches) as determined by the attending anesthesiologist.
  The TOF-Cuff was compared with electromyography
Period: Overall Study
Arm/Group | Moderate Neuromuscular Block, Normal Body Mass Index | Deep Neuromuscular Block, Normal Body Mass Index | Moderate Neuromuscular Block, High Body Mass Index | Deep Neuromuscular Block, High Body Mass Index
Started | 126 | 74 | 43 | 7
Completed | 126 | 74 | 43 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Depth of neuromuscular blockade varied in this observational study. In the Leiden University Medical Centre 148 patients received a moderate neuromuscular blockade whilst 52 received a deep neuromuscular blockade; total 200 patients. In the Dutch Obesity Clinic 21 patients received a moderate neuromuscular blockade whilst 29 received a deep neuromuscular blockade; total 50 patients.
Groups:
- Moderate Neuromuscular Block, Normal Body Mass Index: Patients recruited in the Leiden University Medical Centre with a normal body mass index (18-30) Train of four ratios are collected during moderate neuromuscular blockade.
- Deep Neuromuscular Block, Normal Body Mass Index: Patients recruited in the Leiden University Medical Centre with a normal body mass index (18-30) Post tetanic counts are collected during deep neuromuscular blockade
- Moderate Neuromuscular Block, High Body Mass Index: Measurements during deep neuromuscular block in Patients recruited in the Dutch Obesity Clinic with a high body mass index (>30) Train of four ratios are collected during moderate neuromuscular blockade.
- Deep Neuromuscular Block, High Body Mass Index: Measurements during deep neuromuscular block in Patients recruited in the Dutch Obesity Clinic with a high body mass index (>30) Post tetanic counts are collected during deep neuromuscular blockade
- Total: Total of all reporting groups
Arm/Group | Moderate Neuromuscular Block, Normal Body Mass Index | Deep Neuromuscular Block, Normal Body Mass Index | Moderate Neuromuscular Block, High Body Mass Index | Deep Neuromuscular Block, High Body Mass Index | Total
Number analyzed (Participants) | 148 | 52 | 21 | 29 | 250
Age, Continuous [Median (Full Range); unit: years] — Age in years, see below
  years | 57 [20 to 82] | 51 [19 to 83] | 45 [25 to 65] | 47 [23 to 64] | 55 [19 to 83]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex: either male or female
  Participants
    Female | 86 | 25 | 12 | 23 | 146
    Male | 62 | 27 | 9 | 6 | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Count of participants [Count of Participants; unit: Participants] | 148 | 52 | 21 | 29 | 250

OUTCOME MEASURES:

1. Primary Outcome: Depth of Neuromuscular Block During Moderate Neuromuscular Blockade (Outcome Measure/Row Title Train of Four Ratio) and During Deep Neuromuscular Blockade (Outcome Measure/ Row Title Post Tetanic Count)
Description: Depth of as neuromuscular block will be compared between the Tof-Cuff and electromography at five minute intervals during moderate neuromuscular blockade. Bland-Altman analysis modified for repeated measurements (http://sec.lumc.nl/method_agreement_analysis). This Bland-Altman analysis corrects for between subject variability of repeated paired measurements in individual subjects. Bland-Altman analysis estimates bias and limits of agreement (95% differences between compared devices) between Tof-Cuff and electromography and evaluates instrumental imprecision by calculating the repeatability coefficient, which is equal to the standard deviation of the within-subject variability of each device. For interpretation of the Bland-Altman bias during offset of neuromuscular blockade one can assume that a bias above zero indicates that TOF-Cuff overestimates neuromuscular blockade recovery whilst a bias below zero indicates that Tof-Cuff underestimates neuromuscular blockade recovery.
Time Frame: at 5 minute intervals during the length of the entire procedure [which lasted between 20 to 372 minutes]; a mean of the differences between the TOF-Cuff and electromyography of all measurements is calculated and reported below
Population: The outcome measurement data indicates the difference between both devices (TOF-Cuff versus electromography) of either train of four measurements or post tetanic count measurements . Bias is a unitless number and therefore the number option is chosen as measurement type. It is neither a ratio, median or mean. The bias is zero when there is no difference between measurements.
Measure: Number (95% Confidence Interval); unit: bias
Arm/Group | Moderate Neuromuscular Block, Normal Body Mass Index | Deep Neuromuscular Block, Normal Body Mass Index | Moderate Neuromuscular Block, High Body Mass Index | Deep Neuromuscular Block, High Body Mass Index
Number analyzed (Participants) | 148 | 52 | 21 | 29
bias
  "train-of-four ratio": number analyzed (Participants) | 148 | 0 | 21 | 0
  "train-of-four ratio" | 0.312 [0.287 to 0.338] |  | 0.384 [0.299 to 0.469] |
  "post-tetanic-count": number analyzed (Participants) | 0 | 52 | 0 | 29
  "post-tetanic-count" |  | 3.405 [2.294 to 4.517] |  | -0.17 [-2.872 to 2.531]
Statistical Analysis 1: Comparison: Moderate Neuromuscular Block, Normal Body Mass Index vs Moderate Neuromuscular Block, High Body Mass Index; Paired measurements were compared using a Bland-Altman analysis modified for repeated measurements (http://sec.lumc.nl/method_agreement_analysis, Leiden, the Netherlands). This Bland-Altman analysis corrects for between subject variability of repeated paired measurements in individual subjects; Test type: Other — Bland-Altman analysis estimates bias between TOF-Cuff and electromyography; bias = 0.0, 0.05% CI 2-sided [-0.05 to 0.05]

ADVERSE EVENTS:
Time Frame: One month postoperative collection of (serious) adverse event conform the definition of clinicaltrials.gov
Arm/Group | Moderate Neuromuscular Block, Normal Body Mass Index | Deep Neuromuscular Block, Normal Body Mass Index | Moderate Neuromuscular Block, High Body Mass Index | Deep Neuromuscular Block, High Body Mass Index
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/52 | 0/21 | 0/29
Serious Adverse Events (participants affected / at risk) | 7/148 | 3/52 | 0/21 | 0/29
Other Adverse Events (participants affected / at risk) | 13/148 | 7/52 | 0/21 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Neuromuscular Block, Normal Body Mass Index (N=148) | Deep Neuromuscular Block, Normal Body Mass Index (N=52) | Moderate Neuromuscular Block, High Body Mass Index (N=21) | Deep Neuromuscular Block, High Body Mass Index (N=29)
Postoperative prolonged hospital admission (Injury, poisoning and procedural complications) | 7 (7) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Neuromuscular Block, Normal Body Mass Index (N=148) | Deep Neuromuscular Block, Normal Body Mass Index (N=52) | Moderate Neuromuscular Block, High Body Mass Index (N=21) | Deep Neuromuscular Block, High Body Mass Index (N=29)
Postoperative procedural complications (Injury, poisoning and procedural complications) | 13 (13) | 7 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT03117387/Prot_SAP_000.pdf